CLINICAL TRIAL: NCT05308147
Title: Determination of the Postprandial Glycemic Response and Glycemic Index of Nutritional Products: A Randomized Controlled Clinical Trial in Healthy Individuals (v2.0)
Brief Title: Assessment of the Glycemic Responses to Nutritional Products (v2.0)
Acronym: GLIN#2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: INQ-2137 v2.0
Record Dates: First submitted 2022-03-11; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Glycemic Response
Keywords: Glycemic response; Glycemic index; Nutritional products; Healthy individuals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Reference) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: First Reference product
- Arm 2 (Reference) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Second Reference product
- Arm 3 (Reference) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Third Reference product
- Arm 4 (Concept) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: First Concept product
- Arm 5 (Concept) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Second Concept product
- Arm 6 (Concept) (Other): All subjects will receive all interventions during the trial. The order of the Nutritional products will be randomized.
  Interventions: Dietary Supplement: Third Concept product

INTERVENTIONS:
Dietary Supplement: First Reference product — Dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 1 (Reference)
Dietary Supplement: Second Reference product — Dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 2 (Reference)
Dietary Supplement: Third Reference product — Dextrose (containing 25 grams of carbohydrates)
  Arms: Arm 3 (Reference)
Dietary Supplement: First Concept product — Infant Formula (containing 25 grams of carbohydrates)
  Arms: Arm 4 (Concept)
Dietary Supplement: Second Concept product — Infant Formula with new carbohydrate mixture 1 (containing 25 grams of carbohydrates)
  Arms: Arm 5 (Concept)
Dietary Supplement: Third Concept product — Infant Formula with new carbohydrate mixture 2 (containing 25 grams of carbohydrates)
  Arms: Arm 6 (Concept)

SUMMARY:
This study assesses the glycemic responses to nutritional products. During a study visit fasted subjects will consume one serving of the reference product or the test product. Capillary blood samples will be taken at baseline and at several time-points over a 2-hr period. Several nutritional products will be tested over time.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65 years
* Body mass index (BMI) between 18.5 and 27 kg/m²

Exclusion Criteria:

* Known history of gastrointestinal disease, bariatric surgery, AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), or any condition which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2)affect the results.
* Use of medications known to influence carbohydrate metabolism, gastrointestinal function or appetite, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or any medication which might, in the opinion of the medical director either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Known intolerance, sensitivity or allergy to test products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc.).
* History of cancer in the prior two years, except for non-melanoma skin cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
The glycemic index of nutritional products | 3 months

SECONDARY OUTCOMES:
The postprandial glucose levels at each time point after each test product compared with the mean of the 3 references | 3 months
The postprandial incremental area under the curve (iAUC) after each test product compared with the mean of the 3 references | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- INQUIS Clinical Research, Ltd, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No